CLINICAL TRIAL: NCT01017978
Title: Quantitative MR Biomarkers for Sarcoma Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Gary Luker M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HUM 00023415
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Soft Tissue Tumors
MeSH Terms: conditions — Soft Tissue Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI Scan (Other): MRI scan of soft tissue tumor
  Interventions: Procedure: MRI Scan of soft tissue tumor

INTERVENTIONS:
Procedure: MRI Scan of soft tissue tumor — MRI scan will be completed at baseline (prior to start of subject's clinically ordered chemotherapy treatments.

SUMMARY:
To determine if MRI imaging can be used to accurately determine if a sarcoma is responding to the type of chemotherapy being used.

DETAILED DESCRIPTION:
The purpose of this study is to determine if MRI imaging can be used to accurately determine if a sarcoma is responding to the type of chemotherapy being used or if it is ineffective early on in the treatment; instead of finding this out 2-3 months later. If it is determined that MRI can accurately diagnose tumor response, medications can be switched early on potentially improv8ing the patients'chances of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven primary bone or soft tissue tumor
2. No previous treatment for this malignancy
3. Will be given chemotherapy before having surgery or radiation on the tumor.
4. Are able to undergo a MRI examination
5. If your tumor measures at least 1/2 inch in length.

Exclusion Criteria:

1. Younger than 3 yrs. of age or need general anesthesia(sedation that puts you to sleep) to have a MRI performed.
2. History of Renal Failure
3. Are not able to have a MRI performed for any reason such as you have a pacemaker or other implanted device that may malfunction or move because of the magnetic field inside the MRI room and scanner.
4. Have any history of an allergic reaction to gadolinium based contrast agents (a medication injected in a vein that helps create clearer MRI images.

   -

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine if MRI imaging can accurately determine if a sarcoma (tumor)is responding to the type of chemotherapy being used. | Baseline prior to chemo
  To image and evaluate the size of the soft tissue tumor prior to chemotherapy treatment.

SECONDARY OUTCOMES:
MRI Scan | 3 weeks post start of chemo and end of chemo
  To evaluate the size of the soft tissue tumor after start of chemotherapy to determine if the chemo is having any notable effect on tumor prior to surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Luker, M.D., Principal Investigator — Universityof Michigan Health Systems
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States